CLINICAL TRIAL: NCT07076784
Title: A Study for Evaluating the Effect and Safety of Icariin for Acne and Acne Scars
Brief Title: Topical Icariin on Acne and Acne Scars
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Dae Hun Suh, Principal Investigator, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNUH-ICARIIN
Record Dates: First submitted 2025-07-16; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Acne; Acne Scars
Keywords: Icariin
MeSH Terms: conditions — Acne Vulgaris | interventions — icariin

STUDY DESIGN:
Intervention Model Description: Split-face study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Icariin (Experimental): 3% icariin
  Interventions: Drug: Icariin
- Control (Placebo Comparator): 3% ethanol
  Interventions: Drug: Vehicle Control

INTERVENTIONS:
Drug: Icariin — Topical application of 3% icariin solution
  Arms: Icariin
Drug: Vehicle Control — Topical application of 3% ethanol solution
  Arms: Control

SUMMARY:
The goal of this clinical trial is to examine whether topical application of icariin can improve acne and atrophic acne scars in adults. The main questions it aims to answer are:

* Does icariin reduce the number of facial acne lesions and acne scars?
* What histological changes occur in acne or scar tissue after using icariin? Researchers will compare icariin to a vehicle control (3% ethanol solution) to assess its relative efficacy.

Participants will:

* Apply icariin or control solution to each side of the face twice daily for 2 months
* Visit the clinic every 4 weeks for checkup
* Receive skin biopsies before and after the study period, if they consent to this procedure

DETAILED DESCRIPTION:
Acne vulgaris is one of the most common dermatologic conditions, affecting more than 80-90% of adolescents worldwide. Its pathogenesis is multifactorial, involving excessive sebum production, follicular hyperkeratinization, proliferation of Cutibacterium acnes, and inflammation. Clinical manifestations range from comedones and papules to pustules and nodules, most frequently appearing on the face. Beyond the physical burden, facial acne induces significant psychosocial distress, including anxiety, depression, and social withdrawal. Inflammatory lesions frequently progress to atrophic scars, which persist long term and further intensify psychological morbidity. Studies report acne scarring in up to 95% of patients, with approximately 30% developing scars that are severe enough to require clinical intervention.

Current treatments for atrophic acne scars-such as laser resurfacing, chemical peels, microneedling, and soft-tissue fillers-entail risks including pain, prolonged downtime, and variable efficacy. Topical pharmacologic agents, including retinoids, offer noninvasive alternatives, but their scar-remodeling effects are limited and may cause irritation or photosensitivity. Because scar formation involves a complex interplay of inflammation, collagen degradation, and impaired wound healing, there remains an unmet need for therapies that are safe, effective, and accessible, capable of addressing both active acne and established scars.

Icariin is a prenylated flavonoid glycoside isolated from Epimedium species (e.g., Yin Yang Huo, horny goat weed), traditionally used in oriental medicine as an herbal remedy and dietary tincture. It has demonstrated neuroprotective, cardiovascular, anti-osteoporotic, and antitumor effects, and is considered safe for human consumption. Preclinical evidence indicates that icariin inhibits inflammation, regulates lipid metabolism, suppresses bacterial proliferation, and promotes skin wound healing. Despite these properties, which suggest both anti-acne and pro-remodeling potential, no clinical study to date has evaluated icariin's efficacy in human acne or acne scars.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 to 39 with inflammatory acne and atrophic acne scars on both sides of the face

Exclusion Criteria:

* Diagnosis of acne conglobata or acne fulminans
* Pregnancy or breastfeeding
* Presence of systemic diseases or use of medications that may affect acne or scarring
* Presence of psychiatric disorders
* Recent use of isotretinoin within the past 4 months
* Use of other oral or topical acne treatments or anti-acne cosmetics within the past 2 weeks
* Receipt of procedural treatment for acne scars (e.g. chemical peels or energy-based devices) within the past 4 weeks

Ages: 19 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the total number of acne lesions and scars at 8 weeks | From enrollment to the end of treatment at 8 weeks

SECONDARY OUTCOMES:
Investigator's global assessment for acne (IGA) | From enrollment to the end of treatment at 8 weeks
Scar global assessment (SGA) | From enrollment to the end of treatment at 8 weeks
Change from baseline in ECCA scar grading scale at 8 weeks | From enrollment to the end of treatment at 8 weeks
  The ECCA grading scale (échelle d'évaluation clinique des cicatrices d'acné; a French acronym that translates to Clinical Evaluation Scale for Acne Scars in English) is a tool designed to help dermatologists to assess the severity of acne scars. This score ranges from 0 to 540, with higher scores indicating a more severe condition.
Change from baseline in the number of acne lesions and scars by size and type at 8 weeks | From enrollment to the end of treatment at 8 weeks
  Acne lesions by type (inflammatory and noninflammatory); acne scars by size (small-sized, < 2 mm; medium-sized, 2-4 mm; large-sized, > 4 mm) and type (icepick, boxcar, and rolling)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea